CLINICAL TRIAL: NCT04469231
Title: A Multi-Center, Prospective, Historically Controlled Pivotal Trial Comparing The Safety And Effectiveness Of The Synergy Disc To Anterior Cervical Discectomy And Fusion In Patients With One-Level Symptomatic Cervical Degenerative Disc Disease (DDD).
Brief Title: The Synergy Disc To Anterior Cervical Discectomy and Fusion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synergy Spine Solutions (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110-00001
Record Dates: First submitted 2020-07-07; First posted 2020-07-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cervical Degenerative Disc Disease

STUDY DESIGN:
Intervention Model Description: A multicenter, prospective, non-randomized, historically controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Synergy Disc (Experimental): The Synergy Disc is a cervical disc prosthesis that can be inserted between C3-C7 in skeletally mature patients after anterior discectomy to provide restoration of motion to the functional spinal unit. The Synergy Disc is designed to restoring kinematics to the cervical spine. The Synergy Disc is intended for use in the cervical spine for reconstruction of the disc following a single level discectomy for intractable radiculopathy and/or myelopathy.
  Interventions: Device: Anterior Cervical Discectomy & Fusion

INTERVENTIONS:
Device: Anterior Cervical Discectomy & Fusion — ACDF
  Other Names: ACDF

SUMMARY:
A multicenter, prospective, non-randomized, historically controlled study. Demonstrate the Synergy Disc is at least as safe and effective as conventional anterior cervical discectomy and fusion (ACDF) to treat cervical degenerative disc disease (DDD) in subjects who are symptomatic at only one level from C3 to C7 that are unresponsive to conservative management. Patients will be evaluated preoperatively, at the time of surgery, and at 6 weeks, 3, 6, 12, and 24 months after surgery. Follow-up will continue annually until the last patient reaches 24-month follow-up. The primary analysis will occur at 24 months.

DETAILED DESCRIPTION:
The proposed investigation is a prospective, non-randomized, multi-center, historically controlled comparison of the Synergy Disc to the control of conventional anterior cervical discectomy and fusion (ACDF) surgery in patients with cervical DDD. A total of 175 patients will be enrolled to the investigational group. The investigational group results will be compared to a historical control data from the ACDF control group, which utilized an identical study design. A statistically rigorous observational study design using propensity score (PS) subclassification will be used to demonstrate covariate balance and enhance the quality of inferences regarding effectiveness and safety relative to ACDF control. After investigational device enrollment is complete, but before most investigational device subjects have reached their 24-month endpoint, a data set containing only baseline covariates of prospectively enrolled investigational device patients and historical ACDF control patients will be constructed. The propensity score methods detailed below will be implemented by an outcomes-blinded statistician. A Propensity Score Memo summarizing the proposed observational design will be developed and submitted for review by stakeholders including FDA. The outcomes-blinded statistician will remain blinded until after consensus is achieved that the design is acceptable. This will allow for additional outcomes-blinded PS modeling if required. The objective of this clinical trial is to demonstrate the Synergy Disc is at least as safe and effective as conventional ACDF to treat cervical DDD in subjects who are symptomatic at only one level from C3 to C7 that are unresponsive to conservative management.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 70 years;
2. Diagnosis of radiculopathy or myelopathy of the cervical spine, with either radiculopathy symptoms - pain, paresthesia, or paralysis in a specific nerve root distribution C4, C5, C6, or C7, including at least one of the following: arm/shoulder pain (at least 30 mm on 100 mm VAS scale); decreased muscle strength of at least one level on the 0-5 scale described below; abnormal sensation, including hyperesthesia or hypoesthesia; and/or abnormal reflexes; or myelopathy symptoms including positive Romberg evaluation, abnormal heel/toe walk, pathologic hyperreflexia or clonus in lower extremity, positive Babinski, or positive Hoffman's;
3. Symptomatic at only one level from C3-C4 to C6-C7;
4. Radiographically determined pathology at level to be treated correlating to primary symptoms, including at least one of the following:

   1. Decreased disc height compared to adjacent levels on radiographic film, CT, or MRI
   2. Degenerative spondylosis on CT or MRI
   3. Disc herniation on CT or MRI.
5. Neck Disability Index (NDI) score ≥ 30/100;
6. Unresponsive to non-operative treatment for six weeks, or has the presence of progressive symptoms or signs of nerve root/spinal cord compression in the face of conservative treatment;
7. Appropriate for treatment using an anterior surgical approach, including having no more than one previous anterior surgical approach to the cervical spine;
8. Ability and willingness to comply with follow-up regimen; and
9. Written informed consent given by subject or subject's legally authorized representative.

Exclusion Criteria:

1. Infection at the site of surgery;
2. History of, or anticipated treatment for, active systemic infection, including HIV infection or hepatitis C;
3. Prior attempted or completed cervical spine surgery, except (1) laminoforaminotomy (greater than 6 months prior to scheduled surgical treatment), which includes removal of disc material necessary to perform a nerve root decompression, with less than one-third facetectomy at any level, or (2) a successful single-level anterior cervical fusion (greater than 6 months prior to scheduled surgical treatment);
4. More than one immobile vertebral level between C1-T1 from any cause, including but not limited to congenital abnormalities, osteoarthritic "spontaneous" fusions, and prior cervical spinal fusions;
5. Previous trauma to the C3-T1 levels resulting in significant bony or disco-ligamentous cervical spine injury;
6. Axial neck pain in the absence of other symptoms of radiculopathy or myelopathy justifying the need for surgical intervention;
7. Radiographic confirmation of severe facet joint disease or degeneration.
8. Osteoporosis: A screening questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation) for females or MORES (Male Osteoporosis Risk Estimation Score), will be used to screen patients to determine those patients who require a Hip DXA, a bone mineral density measurement. A SCORE or MORES ≥ 6 requires a DXA. If DXA is required, exclusion will be defined as a DXA bone density measured T score ≤ -2.5 (The World Health Organization definition of osteoporosis). DXA scans within the last 6 months prior to surgical treatment may be used;
9. Paget's disease, osteomalacia, or any other metabolic bone disease (excluding osteoporosis which is addressed above);
10. Severe diabetes mellitus requiring daily insulin management;
11. Active malignancy: a history of any invasive malignancy (except non-melanoma skin cancer), unless the patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years;
12. Tumor as source of symptoms;
13. Symptomatic DDD or significant cervical spondylosis at two or more levels;
14. Marked cervical instability on resting lateral or flexion/extension radiographs demonstrated by:

    1. Translation > 3.5 mm and/or
    2. 11° angular difference to that of either adjacent level;
15. Known or suspected allergy to cobalt, chromium, molybdenum, titanium, or polyethylene;
16. Severe myelopathy to the extent that the patient is wheelchair bound;
17. Congenital canal stenosis resulting in a canal diameter of < 10 mm, as measured by CT or MRI;
18. Kyphotic segmental angulation of greater than 11 degrees at treatment or adjacent levels;
19. Arachnoiditis;
20. Pregnant (verified in patients of childbearing potential by a negative urine pregnancy test when pre-admission testing is obtained), or interested in becoming pregnant during the duration of the study;
21. Autoimmune disorders that impact the musculoskeletal system (e.g., lupus, rheumatoid arthritis; ankylosing spondylitis);
22. Congenital bony and/or spinal cord abnormalities that affect spinal stability;
23. Spinal axis disease (thoracic or lumbar) to the extent that surgical consideration is likely anticipated within 6 months after the cervical procedure;
24. Other degenerative joint disease (e.g. shoulder, hip, knee) to the extent that surgical consideration is likely anticipated within 6 months after the cervical procedure;
25. Diseases or conditions that would preclude accurate clinical evaluation (e.g. neuromuscular disorders such as diffuse idiopathic skeletal hyperostosis (DISH));
26. Medications that could interfere with fusion or other bone/soft tissue healing (e.g. anticipated continued use of systemic steroid medication postoperatively);
27. Currently experiencing acute episode of major mental illness (psychosis, major affective disorder, or schizophrenia), or manifesting physical symptoms without a diagnosable medical condition to account for the symptoms, which may indicate symptoms of psychological rather than physical origin;
28. Current or recent history of substance abuse (drug or alcohol) per site PI's determination;
29. Morbid obesity, defined as body mass index ("BMI") > 40;
30. Currently using, or planning to use, bone growth stimulators in the cervical spine;
31. Use of any other investigational drug or medical device within the last 30 days prior to surgery;
32. Currently a prisoner;
33. Currently pursuing personal litigation (defined as litigation that will likely influence the patient's ability or willingness to accurately report their treatment outcomes) related to the neck or cervical spine injury; however, involvement in worker's compensation related litigation is not a required exclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
NDI | 24 Month
  ≥ 15-point improvement in NDI Score (out of 100) in subjects at 24 months compared with baseline
Neurological Assessment | 24 Month
  Maintenance or improvement in neurological status (motor and sensory only) at 24 months compared to baseline
SSI | 24 Month
  No study failure due to secondary surgical interventions (revision, removal, re-operation, supplemental fixation) at the index level
Device Related AE | 24 Month
  Absence of major device related adverse events defined as radiographic failure, neurological failure, or failure by adverse event as adjudicated by the CEC.

SECONDARY OUTCOMES:
SF-3 | 6 Week, 3, 6, 12, and 24 Month
  Health Survey (SF-36) at baseline and at each follow-up time-point
VAS | 6 Week, 3, 6, 12, and 24 Month
  Visual analogue scale (VAS) will be used to evaluate pain where a change of at least 20mm will be considered clinically significant. Neck pain as measured on a 100mm VAS at baseline and at each follow-up time-point. Left and Right arm/shoulder pain as measured on a 100mm VAS at baseline and at each follow-up time-point. Please note, this assessment will include a "Worst" to pool together the left or right arm/shoulder scores with the higher baseline score. VAS Hoarseness on a 100mm scale.
Patient Satisfaction | 6 Week, 3, 6, 12, and 24 Month
  Patient Satisfaction Questionnaire
BZ Score | 6 Week, 3, 6, 12, and 24 Month
  Bazaz Dysphagia Score at 24 months compared to baseline
Odom's Criteria | 6 Week, 3, 6, 12, and 24 Month
  Results at 24 months for the investigational Synergy Disc and at 24 months for the control ACDF will also be categorized by the physician according to Odom's Criteria.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Barrow Brain and Spine, Phoenix, Arizona
  - HonorHealth Research Institute/Barrow Brain and Spine, Scottsdale, Arizona
  - Todd H. Lanman, M.D., Beverly Hills, California
  - Orthopedic Specialty Institute, Orange, California
  - Institute of Neuro Innovation, Santa Monica, California
  - Anschutz Medical Center, Aurora, Colorado
  - Kennedy White Orthopaedic Center, Sarasota, Florida
  - Indiana Spine Group, Carmel, Indiana
  - Michigan Orthopedic Surgeons (2), Southfield, Michigan
  - Michigan Orthopedic Surgeons, Southfield, Michigan
  - Upstate Medical University, East Syracuse, New York
  - Hospital for Special Surgery, New York, New York
  - Exiamia EquiHealth, Durham, North Carolina
  - Summit Spine, Portland, Oregon
  - Center for Sports Medicine and Orthopaedic Surgery (CSMO), Chattanooga, Tennessee
  - Central Texas Brain & Spine, Austin, Texas
  - Austin Neurosurgeons, Austin, Texas
  - Texas Spine Care Center, San Antonio, Texas
  - The Disc Replacement Center, West Jordan, Utah
  - Atlantic Brain & Spine, Reston, Virginia